CLINICAL TRIAL: NCT06085378
Title: Efficacy and Safety of Urinary Kallidinogenase in the Treatment of Acute Ischemic Stroke Combined With Type 2 Diabetes Mellitus (TK-SEEK): a Prospective, Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Study
Brief Title: Efficacy and Safety of Urinary Kallidinogenase in the Treatment of Acute Ischemic Stroke Combined With Type 2 Diabetes Mellitus
Acronym: TK-SEEK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-2023-509
Record Dates: First submitted 2023-09-07; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke; Type 2 Diabetes
MeSH Terms: conditions — Ischemic Stroke; Diabetes Mellitus, Type 2 | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary Kallidinogenase for injection (Experimental): Patients in this arm will be given urinary kallidinogenase for injection, 0.15 peptide nucleic acids(PNA), once a day for 10 days
  Interventions: Drug: Urinary Kallidinogenase for injection
- Placebo (Placebo Comparator): An inactive substance identical in appearance to the urinary kallidinogenase for injection, once a day for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Urinary Kallidinogenase for injection — The 0.15 peptide nucleic acids(PNA) unit of Eurecrine for injection was dissolved in 100ml sodium chloride injection by intravenous infusion for not less than 50 minutes, once a day. The solvent can be increased and/or slowed down according to the patient's condition for 10 consecutive days, while receiving clinical routine treatment for 10 days
  Other Names: KLK、HUK
  Arms: Urinary Kallidinogenase for injection
Other: Placebo — The 0.15 peptide nucleic acids(PNA) unit of placebo was dissolved in 100ml sodium chloride injection by intravenous infusion for not less than 50 minutes, once a day. The solvent can be increased and/or slowed down according to the patient's condition for 10 consecutive days, while receiving clinical routine treatment for 10 days.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo parallel control study, aim to evaluate the efficacy and safety of human urinary kallidinogenase in the treatment of acute ischemic stroke with type 2 diabetes.

DETAILED DESCRIPTION:
The study process lasts for a total of 90 days, including the screening period, intervention period, and follow-up period. During the intervention period, the experimental group is treated with Urinary Kallidinogenase, while the control group is treated with placebo for 10 days. Both groups receive routine clinical treatment. All patients are followed up until the 90th day after stroke. The sample size of the study is 630 patients. The ratio of the experimental group to the control group is 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤80 years old;
* Patients with acute ischemic stroke diagnosed with complete anterior circulation infarction (TACI) and partial anterior circulation infarction (PACI) according to Oxfordshire Community Stroke Project classification (OCSP), see Appendix 6;
* Refer to the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes (2020 edition), have been diagnosed with type 2 diabetes (need to have a medical history to confirm), see Appendix 7;
* The time from the occurrence of the stroke to the time of admission is less than 48h. If the exact time of onset is unknown, the time of onset of the patient is defined as "the time that finally seems normal";
* First-ever ischemic stroke or have history of ischemic stroke but mRS≤1 before onset;
* 6≤NIHSS≤20;
* Have provided signed written informed consent from the patient or the patient's legal representative

Exclusion Criteria:

* Acute intracranial hemorrhagic diseases confirmed by imaging: parenchymal hemorrhage, epidural hematoma, subdural hematoma, ventricle hemorrhage, subarachnoid hemorrhage, etc.
* Patients who are ready to undergo or have undergone intravascular interventional therapy after the onset of the disease;
* Patients who are ready to undergo or have undergone intravenous thrombolytic therapy after the onset of the disease;
* Severe disturbance of consciousness: NIHSS 1a consciousness level score ≥2;
* Patients with fracture, claudication and other factors affecting functional outcome score upon admission;
* After the onset of the disease, Edaravone injection, Edaravone and Dexborneol concentrated solution for injection, Butylphthalide and sodium chloride injection or Butylphthalide soft capsules have been used;
* Chinese patent medicine injection for improving cerebral blood circulation has been applied after the onset of this disease (see 8.4.2 for details);
* Patients with hypotension (blood pressure less than 90/60mmHg) upon admission;
* Have a history of severe food or drug allergy, or have been allergic to or intolerant of Eurecline injection;
* Eurecline for injection has used angiotensin-converting enzyme inhibitor (ACEI) drugs before taking the drug and has not exceeded 5 half-lives (according to the specific drug instructions);
* Patients who are pregnant or breastfeeding and who plan to become pregnant within 90 days;
* Renal failure or severe renal impairment at the time of screening (creatinine clearance < 30ml/min);
* Liver function impairment: alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2.5 times the upper limit of normal, or other known serious liver diseases such as active infection of acute and chronic hepatitis, cirrhosis, etc.;
* Patients with heart failure (NYHA class III or IV), unstable angina pectoris, acute myocardial infarction, severe arrhythmia, and degree II and III cardiac conduction obstruction within 6 months prior to randomization;
* Those who meet the heavy drinking standard in the three months before the screening period, that is, drinking ≥5 standard drinks per day (1 standard drink is equivalent to 120ml wine, 360ml beer or 45ml liquor);
* Patients who have abused or become addicted to drugs (narcotics, drugs) in the past year;
* Patients with malignant tumors or severe systemic diseases with an expected survival of less than 90 days;
* Patients with serious mental disorders or dementia who cannot cooperate to complete informed consent and follow-up;
* Participated in any interventional drug or device clinical trials within 3 months prior to screening;
* Patients deemed unsuitable for study participation by the investigator;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with modified rankin scale (mRS) 0-2 scores at 90±7 days | 90±7 days
  The proportion of patients with modified rankin scale (mRS) 0-2 scores at 90±7 days

SECONDARY OUTCOMES:
The proportion of patients with modified rankin scale (mRS) 0-3 scores at 90±7 days | 90±7 days
  The proportion of patients with modified rankin scale (mRS) 0-3 scores at 90±7 days
Distribution of modified rankin scale (mRS) at 90±7 days | 90±7 days
  Distribution of modified rankin scale (mRS) at 90±7 days
Changes of NIHSS from baseline to 10 days | from baseline to day 10
  Changes of NIHSS from baseline to 10 days
Changes of Barthel index from baseline to 90±7 days | from baseline to day 90±7
  Changes of Barthel index from baseline to 90±7 days
Changes of mini-mental state examination (MMSE) from baseline to 90±7 days | from baseline to day 90±7
  Changes of mini-mental state examination (MMSE) from baseline to 90±7 days
Changes of Montreal cognitive assessment (MoCA) from baseline to 90±7 days | from baseline to day 90±7
  Changes of Montreal cognitive assessment (MoCA) from baseline to 90±7 days

OTHER OUTCOMES:
Changes of fasting blood glucose values from baseline to 10 days | from baseline to day 10
  Changes of fasting blood glucose values from baseline to 10 days
Changes of HBA1c from baseline to 90±7 days | from baseline to day 90±7
  Changes of HBA1c from baseline to 90±7 days
Changes of hypersensitive C-reactive protein (hs-CRP) and interleukin-6 (IL-6) | from baseline to day 10
  Changes of hypersensitive C-reactive protein (hs-CRP) and interleukin-6 (IL-6)
Changes of urea nitrogen, creatinine and urinary protein | from baseline to day 10
  Changes of urea nitrogen, creatinine and urinary protein
Stroke recurrence rate within 90 days | 90 days
  Stroke recurrence rate within 90 days
Incidence, severity, and causality of adverse events (AE) and serious adverse events (SAE) during the intervention | during the intervention
  Incidence, severity, and causality of adverse events (AE) and serious adverse events (SAE) during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zeng, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China